CLINICAL TRIAL: NCT03763045
Title: Evaluation of the Effect of Sildenafil in Hemodialysis Patients With Pulmonary Hypertension
Brief Title: Sildenafil in Hemodialysis Patients With Pulmonary Hypertension
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ali Elbraky, Assistant lecturer of Internal Medicine and Nephrology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Med135
Record Dates: First submitted 2018-11-07; First posted 2018-12-04 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Hypertension; Hemodialysis Complication
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Sildenafil 25: Twenty hemodialysis patients will receive a dose of 25mg sildenafil daily for 3 months.
  Sildenafil 50: Twenty hemodialysis patients will receive a dose of 50mg sildenafil daily for 3 months.
  Placebo: Twenty hemodialysis patients will receive a placebo tablet daily for 3 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sildenafil 25 (Experimental): Twenty hemodialysis patients will receive a dose of 25mg sildenafil daily for 3 months.
  Interventions: Drug: Sildenafil
- Sildenafil 50 (Experimental): Twenty hemodialysis patients will receive a dose of 50mg sildenafil daily for 3 months.
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Twenty hemodialysis patients will receive a placebo tablet daily for 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 25 mg: Phosphodiesterase inhibitor to be taken once daily
  Arms: Sildenafil 25
Drug: Sildenafil — Sildenafil 50 mg: Phosphodiesterase inhibitor to be taken once daily
  Arms: Sildenafil 50
Other: Placebo — Placebo tablet.
  Arms: Placebo

SUMMARY:
Sildenafil is a phosphodiesterase inhibitor that can exert a nitric oxide-mediated vasodilation effect, so it's considered one of the preferred agents especially in hypoxia induced pulmonary hypertension, can achieve pulmonary vasodilation by enhancing sustained levels of cyclic guanosine monophosphate (cGMP) and nitric oxide.

Despite the potential burden of pulmonary hypertension in hemodialysis patients, such agent like sildenafil has limited studies about optimum dose, safety and long term efficacy in End stage renal disease patients on hemodialysis with pulmonary hypertension

DETAILED DESCRIPTION:
1- To evaluate the effect of sildenafil on pulmonary artery pressure and right ventricular function in hemodialysis patients with pulmonary hypertension.

1. Primary outcome:

   ● Reduction in estimated Pulmonary Artery pressure value (ePAP) in mmHg via transthoracic Doppler Echocardiography.
2. Secondary outcomes:

   * Detection of safety of sildenafil in hemodialysis patients.
   * Finding out sildenafil's optimum dose for hemodialysis patients with pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18-80 years old.
2. Patients on maintenance hemodialysis for more than six months receiving 3 sessions / week using bicarbonate dialysate with a low flux filter and heparin as anticoagulant.
3. Estimated Pulmonary Artery Pressure (ePAP) ≥35 mmHg via Doppler echocardiography
4. Urea reduction ratio (URR) will be ≥ 60% for all patients.
5. Dry weight will be targeted in each case to achieve edema-free state.
6. Informed consent in accordance with the Declaration of Helsinki.

Exclusion Criteria:

* 1. Current treatment of pulmonary hypertension (prostacyclin analogues, endothelin receptor antagonists or phosphodiesterase inhibitors).

  2-Heart diseases (congestive heart failure, ischemic heart disease, congenital heart disease).

  3- Lung diseases (chronic obstructive pulmonary disease, pulmonary thromboemboli or tumor, interstitial lung diseases, sleep apnea, pulmonary fibrosis, Sarcoidosis).

  4-Systemic diseases (scleroderma, systemic lupus erythematosus, portal hypertension).

  5-Human immunodeficiency virus (HIV) infection. 6-History of hypersensitivity to sildenafil. 7-Treatment with any drugs that may interact with sildenafil (Erythromycin , Azoles, Saquinavir-CYP3A4 inhibitors- , Bosentan - CYP3A4 inducer-Nitrates ) 8- Uncontrolled hypertension 9- Anemia with hemoglobin level <10 g/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-02-16 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Decrease in Pulmonary Artery Pressure | 3 months
  Decrease in ePAP (mmHg) via Doppler echocardiography Systolic right ventricular (or pulmonary artery)

SECONDARY OUTCOMES:
Transthoracic echocardiography | 3 months
  Decrease in Estimated PASP (Pulmonary Artery Systolic Pressure) in (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Tamer W Elsaid, MD, Study Director — Associate Professor of Internal Medicine and Nephrology
Locations (1):
- Ain Shams University Hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided